CLINICAL TRIAL: NCT00898144
Title: Morphometric Diagnosis of Atypical Glandular Lesions Using a Conventional Pap Smear From GOG-0171 Patients (Enrolled by GOG-Japan) With a Cytologic Diagnosis of Atypical Glandular Cells of Unspecified Significance (AGUS)
Brief Title: Study of Pap Smears From Patients Enrolled on Clinical Trial GOG-171
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000600575; GOG-8007
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3; cervical adenocarcinoma; atypical squamous cells of undetermined significance
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia; Atypical Squamous Cells of the Cervix | interventions — Papanicolaou Test

INTERVENTIONS:
Other: Papanicolaou test
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying Pap smears in the laboratory from women with atypical glandular cells of unspecified significance may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at Pap smears from women enrolled on clinical trial GOG-171.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the diagnostic accuracy of using previously reported morphometric criteria for chromatin distribution, shortest distance between nuclei, and/or the ratio of nucleoli area to nucleus area in a conventional Pap smear from patients with a cytologic diagnosis of atypical glandular cells of unspecified significance (AGUS) to predict the presence of significant glandular lesions (i.e., adenocarcinoma in situ [AIS] or invasive cancer) and/or squamous lesions (i.e., cervical intraepithelial neoplasia [CIN2 or CIN3]) of the cervix.

Secondary

* To optimize the diagnostic accuracy of using chromatin distribution, shortest distance between nuclei, and/or the ratio of nucleoli area to nucleus area in a conventional Pap smear from patients with a cytologic diagnosis of AGUS to predict the presence of significant glandular lesions (i.e., AIS or invasive cancer) and/or squamous lesions (i.e., CIN2 or CIN3) of the cervix.

OUTLINE: Previously collected slides from Pap smears of patients enrolled on clinical trial GOG-171 are assessed for nuclear chromatin distribution, the shortest distances between the central points of neighboring cell nuclei, and nucleoli area/nucleus area (N/N) ratio via morphometric analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed atypical glandular cells of unspecified significance

  * Original Pap smear used to define the diagnosis must be available for review
* Previously enrolled by GOG-JAPAN onto clinical trialGOG-171

  * Must have been eligible and evaluable for the primary objective of GOG-171
  * Gave permission to use specimens for future cancer research in GOG-171
* Underwent a loop electrosurgical excision procedure/large loop excision of the transformation zone (LEEP/LLETZ) procedure on clinical trial GOG-171 to determine the presence of cervical intraepithelial neoplasia (CIN-2 or CIN-3), significant glandular lesions (AIS), or invasive cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Presence of CIN-2 or CIN-3, significant glandular lesions (AIS), or invasive cancer as determined by the GOG Central Pathology Review of the loop electrosurgical excision procedure/large loop excision of the transformation zone tissue specimen

SECONDARY OUTCOMES:
Intensity of nuclear chromatin staining and chromatin distribution
Distance between neighboring nuclei
Nucleoli area to nucleus area ratio (N/N)

CONTACTS AND LOCATIONS:
Overall Officials: Tsunehisa Kaku, MD, Study Chair — Kyushu University Hospital; Keiichi Fujiwara, MD, PhD — Saitama Medical University International Medical Center